CLINICAL TRIAL: NCT06942910
Title: A Multicentre, Randomised, Double-blind, Active-Controlled, 2-arm Parallel-group Treatment, Phase II Study to Evaluate the Efficacy, Safety, and Tolerability of Zibotentan/Dapagliflozin Compared to Dapagliflozin Alone in Adult Participants With Chronic Kidney Disease and High Proteinuria
Brief Title: A Study to Investigate the Effects of Zibotentan/Dapagliflozin Combination Compared to Dapagliflozin Alone in Adult Participants With Chronic Kidney Disease and High Proteinuria
Acronym: ZODIAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AZ-RU-00010
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease With High Proteinuria
Keywords: Zibotentan; Nephrology; Dapagliflozin; Sodium-glucose co-transporter 2; sodium-glucose co-transporter 2 inhibitor; Kidney diseases; Endothelin antagonist; High Proteinuria
MeSH Terms: conditions — Kidney Diseases | interventions — ZD4054; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zibotentan/Dapagliflozin dose A or Zibotentan/Dapagliflozin dose B (Experimental): Drug dose is determined based on eGFR values. Participants will receive daily oral dose of zibotentan/dapagliflozin in fixed dose combination.
  Interventions: Drug: Zibotentan/Dapagliflozin
- Dapagliflozin alone (Active Comparator): Participants will receive daily oral dose of dapagliflozin.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Zibotentan/Dapagliflozin — Participants will receive zibotentan/dapagliflozin in fixed-dose combination as per the arms they are randomized to
  Arms: Zibotentan/Dapagliflozin dose A or Zibotentan/Dapagliflozin dose B
Drug: Dapagliflozin — Participants will receive dapagliflozin in fixed-dose combination as per the arms they are randomized to
  Arms: Dapagliflozin alone

SUMMARY:
A Study to Investigate the Effects of Zibotentan/Dapagliflozin Combination Compared to Dapagliflozin Alone in Adult Participants with Chronic Kidney Disease and High Proteinuria (ZODIAC)

DETAILED DESCRIPTION:
This is a Phase II, multicentre, randomised, double-blind, active-controlled, 2-arm parallel group study to evaluate the efficacy, safety, and tolerability of zibotentan and dapagliflozin in FDC compared to dapagliflozin alone, given QD on top of SoC, in adult participants with CKD and high proteinuria, with or without T2DM.

Participants who are not already on SGLT2i at screening will receive a 28 day run in intervention with SGLT2i (dapagliflozin) QD. All participants will undergo a 12-week double-blind period. At the end of the treatment visit, participants will discontinue the blinded study intervention and begin open-label dapagliflozin monotherapy until the conclusion of the 4-week safety follow-up period.

The results of this study will provide clinical data on efficacy and safety of an innovation treatment in the new region (the Russian Federation), which will be an important additional data source for Zibotentan/Dapagliflozin FDC approval process in the Eurasian Economic Union.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of signing the informed consent.
* Diagnosis of CKD with eGFR ≥ 20 and < 90 mL/min/1.73m2 AND UACR > 700 mg/g (> 79 mg/mmol) or UPCR > 1000 mg/g (> 113 mg/mmol).
* Body mass index (BMI) within the range ≤40 kg/m2.
* Female participants must be either - not of child-bearing potential or - women of childbearing potential (WOCBP) using at least one highly effective birth control method for at least 3 months prior to first dose of study intervention.
* All WOCBP must have a negative serum pregnancy test result at screening.
* Receiving RAASi therapy (ACEi or ARB), and for the patient maximum tolerated labelled daily dose, that has been stable for at least 4 weeks.

Exclusion Criteria:

* Clinically significant, unstable, or uncontrolled medical condition which in the Investigator's opinion makes it undesirable for the participant to participate in the study.
* Known hypersensitivity to dapagliflozin or zibotentan or any of the excipients of the investigational product. History or ongoing allergy/hypersensitivity, as judged by the investigator, to SGLT2i therapy or ERAs.
* NYHA class III or class IV HF.
* Participants hospitalised for HF and/or who have not been stable on HF therapy during the last 6 months prior to screening.
* HF due to cardiomyopathies that would primarily require other specific treatment.
* High output HF (eg, due to hyperthyroidism or Paget's disease).
* HF due to primary cardiac valvular disease/dysfunction, severe functional mitral or tricuspid valve insufficiency, or planned cardiac valve repair/replacement.
* Evidence of rales or jugular venous distention on physical examination.
* Type 1 diabetes mellitus.
* History of any life-threatening ventricular dysrhythmia (continuous or paroxysmal).
* Participants hospitalised for heart disease or cardiac procedures or for COVID-19 during the last 3 months prior to screening.
* History of solid organ transplantation or bone marrow transplant.
* Any condition with a life expectancy of less than 1 year based on investigator´s clinical judgment.
* Malignancy within the past 5 years. Exceptions to this criterion include non-melanoma skin cancer and curatively treated cervical carcinoma in situ.
* Significant liver disease as judged by the investigator.
* Renal replacement therapy or previous kidney transplant.
* Known history of significant drug or alcohol abuse within 12 months of screening.
* On treatment with strong or moderate CYP3A4 inducer.
* On systemic immunosuppression therapy other than prespecified stable maintenance therapy.
* Participants treated or expecting to be treated with tolvaptan (including as part of participation in a clinical trial), any other ERAs, or budesonide (where used to treat IBD or IgAN).
* Systolic blood pressure above 160 mmHg and/or below 90 mmHg.
* Significant impairment of liver function defined as AST or ALT >3 x upper limit of normal (ULN) or Total serum bilirubin >2 x ULN (an isolated increase in bilirubin in participants with known Gilbert's syndrome is not a reason for exclusion).
* NT-proBNP ≥ 600 pg/mL (or NT-proBNP ≥ 1200 pg/mL, if associated with atrial fibrillation) measured by local laboratory at screening.
* Any of the following results of echocardiography at screening:

  * left ventricular ejection fraction (LVEF) < 50%
  * significant ventricular wall motion abnormality or severe cardiac valve abnormalities
  * isolated pulmonary arterial hypertension (as defined by local clinical practice) or right ventricular failure; in the absence of left-sided HF
* Women who are pregnant, breast-feeding, or women with intent of getting pregnant.
* Women who are not willing to use adequate contraception or cannot, in the opinion of the Investigator, understand and/or comply with the study requirements regarding contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in log-transformed Urinary Albumin to Creatinine Ratio (UACR) from baseline | At Week 12
  To estimate the efficacy of zibotentan and dapagliflozin in FDC versus dapagliflozin alone in reducing albuminuria

SECONDARY OUTCOMES:
Change in log-transformed Urinary Protein to Creatinine Ratio (UPCR) from baseline | At Week 12
  To estimate the efficacy of zibotentan and dapagliflozin in FDC versus dapagliflozin alone in reducing proteinuria
Change in systolic and diastolic blood pressure (BP) from baseline | At Week 12
  To estimate the efficacy of zibotentan and dapagliflozin in FDC versus dapagliflozin alone in reducing systolic and diastolic BP
Number of participants experiencing adverse events | From Week 1 (Day 1) until Follow-up visit (Week 18, Day 112)
  To assess the safety and tolerability of treatment with zibotentan and dapagliflozin in FDC compared to dapagliflozin alone during 12 weeks of treatment and 4 weeks of safety follow-up

OTHER OUTCOMES:
Change in estimated Glomerular Filtration Rate (eGFR) from baseline | At Week 12
  To explore the effect of zibotentan and dapagliflozin in FDC versus dapagliflozin alone to slow decline in kidney function, as measured by eGFR
Proportion of participants achieving Urine Protein to Creatinine Ratio (UPCR) < 1000 mg/g and > 30% reduction from baseline | Across the visits from Week 2 (Day 14) up to Week 12 (Day 84)
  To explore the effect of zibotentan and dapagliflozin in FDC versus dapagliflozin alone to reduce proteinuria, as measured by the proportion of participants achieving UPCR < 1000 mg/g and > 30% reduction from baseline
Proportion of participants achieving Urinary Albumin to Creatinine Ratio (UACR) < 300 mg/g | Across the visits from Week 2 (Day 14) up to Week 12 (Day 84)
  To explore the effect of zibotentan and dapagliflozin in FDC versus dapagliflozin alone to reduce albuminuria, as measured by the proportion of participants achieving UACR < 300 mg/g

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - Research Site, Aramil
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at : https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home